CLINICAL TRIAL: NCT03900312
Title: Intergenerational Strengths-Based Program for American Indian Girls as They Transition to Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9117
Record Dates: First submitted 2019-02-28; First posted 2019-04-03 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Sexual Activity; Sex; Alcohol Use; Pregnancy; Drug Use
Keywords: Native American; Youth; Young Adult
MeSH Terms: conditions — Sexual Behavior; Coitus; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The program consists of 11 sessions conducted with girls ages 8-11 and their female caregivers. 5 of the 11 sessions will be taught to groups of 8-12 girls and their mothers, and 6 of the sessions will be taught to individual girl/female caregivers' dyads. The mix of group- and home-based lessons is based on findings from the formative phase about preference for certain topics to be taught in groups vs. individual dyads. Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room. Individual dyad sessions will take place in the girls'/female caregivers home or another private place of their choosing such as our local Johns Hopkins offices.
  Interventions: Behavioral: Asdzaan Be'eena' Program

INTERVENTIONS:
Behavioral: Asdzaan Be'eena' Program — The program will consist of 11 sessions conducted with girls ages 8-11 and their female caregivers. 5 of the 11 sessions will be taught to groups of 8-12 girls and their mothers, and 6 of the sessions will be taught to individual girl/female caregivers' dyads. The mix of group- and home-based lessons is based on findings from the formative phase about preference for certain topics to be taught in groups vs. individual dyads. Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room. Individual dyad sessions will take place in the girls'/female caregivers home or another private place of their choosing such as our local Johns Hopkins offices. The program will be conducted over 2.5-3 months with one session occurring every week for 11 weeks.

SUMMARY:
The investigators will conduct a pilot study to assess the acceptability, feasibility, satisfaction, and participant-level outcomes among girls and their mother/female caregiver participating in a preconception health program. The program was developed through an extensive formative phase and is delivered weekly over ~3 months. The investigators will enroll a total of 60 female caregivers and their 8-11 year old daughters/female children to participate in the program and evaluation. Implementation data including acceptability, feasibility and satisfaction will be collected through REDCap and paper assessments completed after each program session and at the completion of the program. Preliminary impact data will be collected through REDCap up to 3 months post-intervention completion.

The aims are as follows:

1. To understand if the preconception health program is feasible and acceptable among young girls and their mothers or female caregivers
2. To explore optimal implementation of the program to inform future research and scale up.
3. To assess preliminary impact of the preconception health program on girls' and caregiver's knowledge, cultural connectedness, caregiver-child relationship, community and school connectedness, coping skills, parenting self-efficacy, depression, quality of life as well as substance use behaviors and intentions and intention about sexual activity.

DETAILED DESCRIPTION:
The investigators will conduct a pilot evaluation to understand the feasibility, acceptability, satisfaction and explore preliminary impacts of a preconception health program. The primary research question is: Is the preconception health program developed through the formative phase of this study acceptable and feasible to girls and caregiver participants? The program aims to improve the overall health and wellbeing of girls and their female caregivers by decreasing and delaying the initiation of substance use and risk behaviors associated with sexual initiation among adolescent girls. A second research question is: does the preconception health program have preliminary impacts on key protective and risk factors related to substance use and risky sexual behavior among girls and their female caregivers?

The Preconception Health Program will consist of 11 sessions conducted with girls ages 8-11 and their female caregivers. 5 of the 11 sessions will be taught to groups of 8-12 girls and their mothers, and 6 of the sessions will be taught to individual girl/female caregivers' dyads. The mix of group- and home-based lessons is based on findings from the formative phase about preference for certain topics to be taught in groups vs. individual dyads. Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room. Individual dyad sessions will take place in the girls'/female caregivers home or another private place of their choosing such as our local Johns Hopkins offices. The program will be conducted over 2.5-3 months with one session occurring every week for 11 weeks. The total program duration is 660-990 minutes.

To adequately assess the primary research question, the investigators will enroll 60 dyads, grouped into three cohorts of 10 dyads each, who will complete satisfaction questionnaires after each of the program sessions and upon completion of the program. To assess preliminary impact on girls' risk for substance use and intention about sexual activity, including cultural connectedness, mother-daughter communication and psychological health and wellbeing, the investigators will deliver an evaluation conducted at baseline, upon completion of the intervention (post-intervention assessment) and 3 months following completion of the intervention (3-month follow-up assessment). The investigators will also assess program impact on female caregivers' substance use, parent-child communication and factors related to the female caregivers' wellbeing through an evaluation conducted at baseline, upon completion of the intervention (post-intervention assessment) and 3 months following completion of the intervention (3-month follow-up assessment).

ELIGIBILITY:
Inclusion Criteria (Caregivers):

* Female > 18 years of age
* Self-identify as Navajo
* Be a caregiver of a girl 8-11 years old who is available to enroll in the study
* Living within 50 miles of the Chinle (Tsaile or Pinon are also included) or Tuba City, Arizona Johns Hopkins program offices
* Willing to participate in the preconception health program
* Willing to complete all implementation and follow-up assessment
* Speaks and reads English
* Not cognitively or visually impaired (able to complete questionnaires)
* Review and sign informed consent

Inclusion Criteria (Child):

* Female, 8-11 years old
* Have a caregiver enrolled in the study
* Living within 50 miles of the Chinle (Tsaile or Pinon are also included) or Tuba City, Arizona Johns Hopkins program offices
* Willing to participate in the preconception health program
* Willing to complete all implementation and follow-up assessments
* Speaks and reads English
* Not cognitively or visually impaired (able to complete questionnaires)
* Review and sign a study assent and have a parent/guardian sign parental permission

Exclusion Criteria (child and caregiver):

* Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, cognitive impairment, etc.)
* Due to potential mobility of foster children, children in foster care are excluded from the study.

Min Age: 8 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Inclusion Criteria (Caregivers):
  * Female > 18 years of age
  * Self-identify as Navajo
  * Be a caregiver of a girl 8-11 years old who is available to enroll in the study
  Inclusion Criteria (Child):
  • Female, 8-11 years old
Enrollment: 65 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Three month change in child cultural knowledge score on knowledge assessment | Baseline and 3 months post implementation
  Investigators will measure change in knowledge from baseline and 3 months post program completion via a 4-question knowledge assessment completed by the child (score 0-100%). A higher score indicates higher (greater) knowledge.
Three month change in caregiver cultural knowledge score on knowledge assessment | Baseline and 3 months post implementation
  Investigators will measure change in knowledge from baseline and 3 months post program completion via a 10-questions knowledge assessment completed by caregivers (score 0-100%). A higher score indicates higher (greater) knowledge.
Three month change in child reported family engagement in Navajo culture assessed by family engagement questionnaire | Baseline and 3 months post implementation
  Family engagement in the Navajo culture will be assessed via a 4- question assessment that is on a 5-point Likert scale (score: 0-20). The assessment was created by the study team. The investigators will look at the change in total score from baseline to 3 months post implementation. A higher score indicates higher (greater) family engagement.
Three month change in caregiver reported family engagement in Navajo cultural assessed family engagement questionnaire | Baseline and 3 months post implementation
  Family engagement in the Navajo culture will be assessed via a 4-question assessment that is on a 5-point Likert scale (score: 0-20). The assessment was created by the study team. The investigators will look at the change in total score from baseline to 3 months post implementation.
Three month change in child reported parent-child communication assessed by parent-child communication questionnaire at 3 | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on girls' and caregivers' communication via a 20-item assessment on a 5-point Likert scale (score: 0-100). The assessment was created by the study team. Investigators will assess the change in child reported caregiver-child communication from baseline to 3 months post program implementation.
  Parental monitoring will be assessed among caregivers only via a 6-question assessment created by Silverberg and Small.
Three month change in caregiver reported parent-child communication assessed by parent-child communication questionnaire | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on girls' and caregivers' communication via a 20-item assessment on a 5- point likert scale (score: 0-100). The assessment was created by the study team. Investigators will assess in caregiver reported caregiver-child communication from baseline to 3 months post program implementation.
Three month change in caregiver reported parental monitoring assessed by parental monitoring questionnaire | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on parental monitoring via a 6-question assessment created by Silverberg and Small. Investigators will look at the change from baseline to 3 months post program implementation in parental monitoring as reported by caregivers via the parental monitoring scale. Parental monitoring will be assessed among caregivers only via a 6-question assessment created by Silverberg and Small. A higher score indicates a higher (better) parental monitoring.
Three month change in child self-esteem on a self-esteem assessment developed by study team | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on child self-esteem via a 4-item assessment on a 5-point Likert scale (score: 0-20). Investigators will assess the change in total score from baseline to 3 months post implementation. A higher score indicates a higher (better) self-esteem.
Three month change in child self-efficacy on a self-efficacy assessment adapted from Muris 2001. | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on child' self-efficacy via a 5-item assessment on a 5-point likert scale (score: 0-25). Investigators will assess the change in the total score from baseline to 3 months post implementation. Higher score=higher (better) selfefficacy Citation for scale: Muris, P. (2001). Self-Efficacy Questionnaire for Children. Journal of Psychopathology and Behavioral Assessment, 23(3), 145-149.
Three month change in child social support on a social support assessment developed by study team. | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on child social support via a 4-item assessment on a 5-point Likert scale (score: 0-20). Investigators will assess the change in total score from baseline to 3 months post implementation. A higher score indicates a higher (more) social support.
Three month change in average score on risky behaviors assessment | Baseline and 3 months post implementation
  The investigators will assess the impact of the Asdzaan Be'eena program on child attitudes related to risky behaviors via a 6-item assessment on a 5-point Likert scale (score: 0-30). Investigators will assess the change in the total score from baseline to 3 months post implementation. A higher score indicates better attitudes (less endorsement of) risk behaviors.
Three month change in child reproductive health knowledge via a reproductive health knowledge questionnaire | Baseline and 3 months post implementation
  Investigators will measure change in knowledge from baseline and 3 months post program completion via a 3-question knowledge assessment completed by the child (score 0-100%). A higher score indicates more knowledge.
Three month change in caregiver reproductive health knowledge via a reproductive health knowledge questionnaire | Baseline and 3 months post implementation
  Investigators will measure change in knowledge from baseline and 3 months post program completion via a 10-questions knowledge assessment completed by the caregivers (score 0-100%). A higher score indicates higher (more) knowledge.
Three month change in caregiver family mastery via the multicultural mastery scale | Baseline and 3 months post implementation
  Investigators will measure family mastery via a 5-item assessment on a 5-point Likert scale (score: 0-25). Change in total score between baseline and 3 months will be utilized to assess program impact.
Three month change in caregiver friend mastery via the multicultural mastery scale | Baseline and 3 months post implementation
  Investigators will measure communal mastery- friends via a 5-item assessment on a 5-point Likert scale (score: 0-25). Change in total score between baseline and 3 months will be utilized to assess program impact. A lower score indicates higher (better) mastery.
Three month change in caregiver self mastery via the multicultural mastery scale | Baseline and 3 months post implementation
  Investigators will measure communal mastery- self via a 5-item assessment on a 5-point likert scale (score: 0-25). Change in total score between baseline and 3 months will be utilized to assess program impact. A lower score indicates higher (better) mastery.
Three month change in parental self-efficacy via the parenting agency questionnaire (Dumka, 1996) | Baseline and 3 months post implementation
  Investigators will measure parenting self-efficacy via a 10-item assessment on a 5-point Likert scale (score: 0-50). Change in total score between baseline and 3 months will be utilized to assess program impact. A higher score indicates a higher (better) self-efficacy.
  Citation: Dumka, L. E., Stoerzinger, H. D., Jackson, K. M., & Roosaa, M. W. (1996). Examination of the cross-cultural and crosslanguage equivalence of the Parenting Self-Agency Measure. Family Relations, 45, 216-222.
Three month change in average score on the PHQ-9 depression screener | Baseline and 3 months post implementation
  Investigators will measure depression via the Patient Health Questionnaire (PHQ-9) a 9-item assessment (Kroenke 2001). Change in total score between baseline and 3 months will be utilized to assess program impact.
  Citation: Kroenke, K., Spitzer, R. L., & Williams, J. B. (2001). The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine, 16(9), 606-613. https:// doi.org/10.1046/j.1525-1497.2001.016009606.x
Three month change in frequency of activities completed together via a parent-child activity assessment | Baseline and 3 months post implementation
  Investigators will measure caregiver and child activities together via a 5-item assessment on a 5-point likert scale completed by the child (score: 0-25). Change in total score between baseline and 3 months will be utilized to assess program impact.
  A higher score indicates more frequent activities with caregiver.
Three month change in percent of children reporting wanting to have a kinaalda | Baseline and 3 months post implementation
  Investigators will measure child's attitude about having a Kinaalda via one question: "Do you want to have a Kinaalda ceremony when you get your period?". Answers include "yes" and "no". Investigators will assess the difference in the number of children who say "yes" at baseline compared to 3 months post implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Chinle, Arizona, United States

IPD SHARING:
Plan to Share IPD: No